CLINICAL TRIAL: NCT02432131
Title: Incidences of Decompression Sickness in SCUBA DIVERs With or Without Patent Foramen Ovale (DIVER-PFO); A Double-blinded, Prospective Cohort Study
Brief Title: Decompression Sickness in Divers With or Without Patent Foramen Ovale
Acronym: DIVER-PFO
Status: Completed | Type: Observational
Sponsor: Sejong General Hospital (Other)
Collaborators: Sejong Research Institute (Unknown)
Responsible Party: Principal Investigator, Hyun Jong Lee, MD, PhD, Sejong General Hospital
Other Study IDs: DIVER-PFO_ver1.1
Record Dates: First submitted 2015-04-28; First posted 2015-05-01 (Estimated); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Foramen Ovale, Patent; Decompression Sickness
MeSH Terms: conditions — Foramen Ovale, Patent; Decompression Sickness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Divers with PFO
- Divers without PFO

SUMMARY:
The investigators will prospectively estimate incidences of decompression sickness in SCUBA divers with or without patent foramen ovale (PFO). All participants will receive transesophageal echocardiogram and transcranial doppler to ascertain whether they get a PFO. Clinical follow up will be undertaken 3 month after transesophageal echocardiographic evaluation, and every 6 month up to 3 years by E-mailing or telephone interview with self-questionnaire report. All decompression sickness (DC) events or DC-like symptoms will be reviewed by a professional diver, who is a medical doctor and member of DAN-AP, and a neurologist.

DETAILED DESCRIPTION:
PFO was defined as transesophageal echocardiographic (TEE) evidence of infused microbubbles in the left atrium within three cardiac cycles after their appearance in the right atrium, at rest or during Valsalva release. If TEE finding will not be conclusive, we will decide the presence or absence of PFO with supplementary transcranial doppler. It will be blinded to participants, physicians and research persons to perform clinical follow-up. It will be not officially recorded, and will be preserved by another research person, who will not contact study participants.

ELIGIBILITY:
Inclusion Criteria:

* Divers who experienced fifty dives per year

Exclusion Criteria:

* Decompression sickness within recent 20 dives
* Previous procedure or surgery for closure of PFO or ASD
* Previous cerebral infarction or hemorrhage
* Previous epilepsy
* Previous angina or myocardial infarction

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recreational or occupational SCUBA (self-contained underwater breathing apparatus) divers
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-05; Primary Completion 2021-02 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
PFO-related decompression sickness | Three years
  Three-year cumulative incidences of cutaneous or neurological decompression sickness, all symptoms requiring recompression chamber therapy, all symptoms developed during ascending or within 30minute after surfacing, or unexplained death within 2 weeks after diving

SECONDARY OUTCOMES:
Cutaneous or neurological decompression sickness | Three years
All symptoms requiring recompression chamber therapy | Three years
All symptoms developed during ascending or within 30minute after surfacing | Three years
Unexplained death within 2 weeks after diving | Three years

CONTACTS AND LOCATIONS:
Locations (1):
- Sejong general hospital, 91-121 Sosa 2-Dong, Sosa-Gu, Bucheon-si, Gyeonggi-do, South Korea